CLINICAL TRIAL: NCT05485779
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose, and Food Effect Evaluation Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of AQ280 in Healthy Subjects
Brief Title: SAD, MAD and Food Effect Evaluation of Safety, Tolerability, and PK of AQ280 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AQILION AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ARIA-1
Record Dates: First submitted 2022-07-15; First posted 2022-08-03 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part A (SAD): Group A1 (Experimental): Single dose of AQ280, 3 mg or placebo
  Interventions: Drug: AQ280; Drug: Placebo
- Part A (SAD): Group A2 (Experimental): Single dose of AQ280, dose to be determined (TBD) or placebo
  Interventions: Drug: AQ280; Drug: Placebo
- Part A (SAD): Group A3 (Experimental): Single dose of AQ280, dose TBD or placebo
  Interventions: Drug: AQ280; Drug: Placebo
- Part A (SAD): Group A4 (Experimental): Single dose of AQ280, dose TBD or placebo
  Interventions: Drug: AQ280; Drug: Placebo
- Part A (SAD): Group A5 (Experimental): Single dose of AQ280, dose TBD or placebo
  Interventions: Drug: AQ280; Drug: Placebo
- Part B (MAD): Group B1 (Experimental): AQ280 dose TBD or placebo, once daily (QD) for seven days
  Interventions: Drug: AQ280; Drug: Placebo
- Part B (MAD): Group B2 (Experimental): AQ280 dose TBD or placebo, once daily (QD) for seven days
  Interventions: Drug: AQ280; Drug: Placebo
- Part B (MAD): Group B3 (Experimental): AQ280 dose TBD or placebo, once daily (QD) for seven days
  Interventions: Drug: AQ280; Drug: Placebo

INTERVENTIONS:
Drug: AQ280 — Dose form: capsule, hard
  Strength: 3 to 100 mg
  Method of administration: oral
Drug: Placebo — Active substance: none
  Dose form: capsule, hard
  Strength/dose: not applicable
  Method of administration: oral

SUMMARY:
The principal aim of this study is to obtain safety and tolerability data when AQ280 is administered orally as single and multiple doses to healthy subjects. This information, together with the pharmacokinetic (PK) data, will help establish the doses and dosing regimen suitable for future studies in patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all of the following criteria at the screening visit (and/or at check-in, where noted):

1. Males or females, of any race, between 18 and 65 years of age, inclusive.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive.
3. In good health, determined by no clinically significant findings from medical history, 12 lead ECG, vital sign measurements, and clinical laboratory evaluations at screening and check-in and from the physical examination at check-in, as assessed by the investigator (or designee).
4. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
5. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.

Exclusion Criteria:

Subjects will be excluded from the study if they satisfy any of the following criteria at the screening visit (or at check-in, where noted):

Medical conditions

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, as determined by the investigator (or designee).
3. History of any surgical (eg, stomach or intestinal surgery or resection) or medical condition that would potentially alter absorption, distribution, metabolism, and/or excretion of orally administered drugs. Uncomplicated appendectomy and hernia repair will be allowed. Cholecystectomy will not be allowed.
4. History of any significant infectious disease, as assessed by the investigator, within 2 weeks prior to the first dose of IMP.
5. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) values >1.2 × upper limit of normal (ULN).
6. Congenital nonhemolytic hyperbilirubinemia (including suspicion of Gilbert's syndrome).
7. Hemoglobin value, neutrophil count, and/or lymphocyte count <lower limit of normal.
8. Clinically significant abnormal ECG at screening or check-in.
9. Positive hepatitis panel and/or positive human immunodeficiency virus test. Subjects whose results are compatible with prior immunization may be included at the discretion of the investigator
10. Current active tuberculosis based on Quantiferon™ tuberculosis Gold test.

    Prior/concomitant therapy
11. Administration of a coronavirus disease 2019 vaccine in the past 30 days prior to the first dose of investigational medicinal product (IMP).
12. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to the first dose of IMP, unless deemed acceptable by the investigator (or designee).
13. Use or intend to use any prescription medications/products other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives within 14 days prior to the first dose of IMP, unless deemed acceptable by the investigator (or designee).
14. Use or intend to use slow release medications/products considered to still be active within 14 days prior to check in, unless deemed acceptable by the investigator (or designee).
15. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 7 days prior to check in, unless deemed acceptable by the investigator (or designee).

    Prior/concurrent clinical study experience
16. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to dosing.
17. Have previously completed or withdrawn from this study.

    Diet and lifestyle
18. Alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
19. Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at screening or check-in.
20. History of alcoholism or drug/chemical abuse within 2 years prior to check-in.
21. Smoking >5 cigarettes per day, on average, or use the equivalent tobacco- or nicotine containing products per day.
22. Ingestion of poppy seed , Seville orange , star fruit-, or grapefruit containing foods or beverages within 7 days prior to check-in.

    Other exclusions
23. Receipt of blood products within 2 months prior to check-in.
24. Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
25. Poor peripheral venous access.
26. Subjects who, in the opinion of the investigator (or designee), should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Törnell, MD, PhD, Study Director — AQILION AB
Locations (1):
- Fortrea Clinical Research Unit Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A (SAD): Placebo (Fasted): Single dose of placebo, fasted
  Dose form: capsule, hard Method of administration: oral
- Part A (SAD): 3 mg (Fasted): Single dose of 3 mg AQ280, fasted
  AQ280: Dose form: capsule, hard Method of administration: oral
- Part A (SAD): 9 mg (Fasted): Single dose of 9 mg AQ280, fasted
  AQ280: Dose form: capsule, hard Method of administration: oral
- Part A (SAD): Placebo (Fasted/Fed): Single dose of placebo fasted on Day 1 of Treatment Period 1 and fed on Day 1 of Treatment Period 2.
  Dose form: capsule, hard Method of administration: oral
- Part A (SAD): 16 mg (Fasted/Fed): Single dose of 16 mg AQ280 fasted on Day 1 of Treatment Period 1 and fed on Day 1 of Treatment Period 2.
  AQ280: Dose form: capsule, hard Method of administration: oral
- Part A (SAD): 48 mg (Fasted): Single dose of 48 mg AQ280, fasted
  AQ280: Dose form: capsule, hard Method of administration: oral
- Part A (SAD): 60 mg (Fasted): Single dose of 60 mg AQ280, fasted
  AQ280: Dose form: capsule, hard Method of administration: oral
- Part B (MAD): Placebo: Placebo, once daily (QD) for seven days
  Dose form: capsule, hard Method of administration: oral
- Part B (MAD): 9 mg: AQ280 9 mg once daily (QD) for seven days
  AQ280: Dose form: capsule, hard Method of administration: oral
- Part B (MAD): 27 mg: AQ280 27 mg once daily (QD) for seven days
  AQ280: Dose form: capsule, hard Method of administration: oral
- Part B (MAD): 60 mg: AQ280 60 mg once daily (QD) for seven days
  AQ280: Dose form: capsule, hard Method of administration: oral
Period: Treatment Period 1 (Fasted)
Arm/Group | Part A (SAD): Placebo (Fasted) | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): Placebo (Fasted/Fed) | Part A (SAD): 16 mg (Fasted/Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted) | Part B (MAD): Placebo | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
Started | 8 | 6 | 6 | 2 | 6 | 6 | 6 | 7 | 7 | 6 | 6
Completed | 8 | 6 | 6 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 2 (Fed Groups Only)
Arm/Group | Part A (SAD): Placebo (Fasted) | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): Placebo (Fasted/Fed) | Part A (SAD): 16 mg (Fasted/Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted) | Part B (MAD): Placebo | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
Started (Fed Groups only in Treatment Period 2) | 0 | 0 | 0 | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Discontinued prior to dosing in fed period due to a failed drug screen at check-in | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A (SAD): Placebo (Fasted) | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): Placebo (Fasted/Fed) | Part A (SAD): 16 mg (Fasted/Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted) | Part B (MAD): Placebo | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 2 | 6 | 6 | 6 | 7 | 7 | 6 | 6 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (11.65) | 38.8 (15.46) | 40.0 (14.70) | 32.0 (7.07) | 53.5 (13.63) | 39.8 (21.78) | 43.0 (18.21) | 38.0 (13.96) | 43.6 (12.75) | 36.3 (14.64) | 47.8 (13.67) | 43.0 (14.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 0 | 1 | 4 | 3 | 1 | 5 | 1 | 3 | 26
  Male | 5 | 3 | 4 | 2 | 5 | 2 | 3 | 6 | 2 | 5 | 3 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 6 | 2 | 6 | 6 | 6 | 7 | 7 | 6 | 6 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
  White | 6 | 6 | 6 | 2 | 6 | 4 | 6 | 7 | 5 | 5 | 5 | 58
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeters] | 172.58 (9.031) | 175.32 (7.802) | 173.48 (11.127) | 180.05 (6.293) | 179.65 (4.281) | 165.20 (10.623) | 170.87 (12.692) | 174.90 (17.240) | 168.37 (6.033) | 172.35 (9.957) | 170.47 (7.277) | 172.54 (10.192)
Body weight [Mean (Standard Deviation); unit: kilograms] | 80.15 (12.279) | 73.88 (12.495) | 83.48 (12.015) | 81.25 (15.486) | 85.20 (8.323) | 62.17 (14.016) | 75.12 (17.688) | 77.77 (15.225) | 65.91 (7.416) | 72.6 (18.304) | 66.73 (11.898) | 74.62 (14.251)
Body mass index [Mean (Standard Deviation); unit: kilograms/meter^2] | 26.90 (3.601) | 23.97 (3.315) | 27.68 (2.218) | 24.95 (3.041) | 26.37 (2.069) | 22.67 (3.647) | 25.55 (4.157) | 25.37 (2.914) | 23.23 (2.319) | 24.15 (4.097) | 22.88 (2.785) | 24.92 (3.369)

OUTCOME MEASURES:

1. Primary Outcome: Part A (SAD): Number of Treatment Emergent Adverse Events (TEAEs) by Participant
Description: The number of participants who experienced a treatment-emergent event (TEAE) are presented.
Time Frame: Part A (SAD): Screening up to Day 8 for fasted cohorts and Day 18(±2) for fed/fasted cohorts
Population: Safety population. The 'Part A (SAD): Placebo (Fasted)' cohort includes the 8 participants in the fasted only cohort as well as any AEs experienced by the 2 participants in the 'Part A (SAD): Placebo (Fasted/Fed)' cohort whilst in the fasting during Treatment Period 1. Any AEs experienced by these 2 participants during Treatment Period 2 (ie, the fed stage) only are listed separately under the cohort 'Part A (SAD): Placebo (Fed).
Measure: Count of Participants; unit: Participants
Groups:
- Part A (SAD): Placebo (Fed): Single dose of placebo, fed
  Dose form: capsule, hard Method of administration: oral
- Part A (SAD): 16 mg (Fasted): Single dose of 16 mg AQ280, fasted
  AQ280: Dose form: capsule, hard Method of administration: oral
- Part A (SAD): 16 mg (Fed): Single dose of 16 mg AQ280, fed
  AQ280: Dose form: capsule, hard Method of administration: oral
Arm/Group | Part A (SAD): Placebo (Fasted) | Part A (SAD): Placebo (Fed) | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): 16 mg (Fasted) | Part A (SAD): 16 mg (Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted)
Number analyzed (Participants) | 10 | 2 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 1

2. Primary Outcome: Part A (SAD): Number of Treatment Emergent Adverse Events (TEAEs) Experienced
Description: The number of total events experienced by participants are presented.
Time Frame: Part A (SAD): Screening up to Day 8 for fasted cohorts and Day 18(±2) for fed/fasted cohorts
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Part A (SAD): Placebo (Fasted) | Part A (SAD): Placebo (Fed) | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): 16 mg (Fasted) | Part A (SAD): 16 mg (Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted)
Number analyzed (Participants) | 10 | 2 | 6 | 6 | 6 | 6 | 6 | 6
events | 1 | 0 | 1 | 2 | 2 | 3 | 0 | 1

3. Primary Outcome: Part B (MAD): Number of Treatment Emergent Adverse Events (TEAEs) by Participant
Description: The number of participants who experienced a treatment-emergent event (TEAE) are presented.
Time Frame: Part B (MAD): Screening up to Day 14(±3)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (MAD): Placebo | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
Number analyzed (Participants) | 7 | 7 | 6 | 6
Participants | 3 | 3 | 3 | 3

4. Primary Outcome: Part B (MAD): Number of Treatment Emergent Adverse Events (TEAEs) Experienced
Description: The number of total TEAE events experienced by participants are presented.
Time Frame: Part B (MAD): Screening up to Day 14(±3)
Population: Safety Population
Measure: Number; unit: events
Arm/Group | Part B (MAD): Placebo | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
Number analyzed (Participants) | 7 | 7 | 6 | 6
events | 7 | 6 | 8 | 4

5. Primary Outcome: Part A (SAD): Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: The number of participants with clinically significant abnormalities in vital signs is presented.
  Vital signs: systolic and diastolic blood pressure, pulse rate, and oral body temperature
Time Frame: Part A (SAD): Screening up to Day 3
Population: Safety population. The 'Part A (SAD): Placebo (Fasted)' cohort includes the 8 participants in the fasted only cohort as well as any results for the 2 participants in the 'Part A (SAD): Placebo (Fasted/Fed)' cohort whilst in the fasting during Treatment Period 1. Results for the 2 participants during Treatment Period 2 (ie, the fed stage) only are listed separately under the cohort 'Part A (SAD): Placebo (Fed)'.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (SAD): Placebo (Fasted) | Part A (SAD): Placebo (Fed) | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): 16 mg (Fasted) | Part A (SAD): 16 mg (Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted)
Number analyzed (Participants) | 10 | 2 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part A (SAD): Number of Participants With Abnormal ECG
Description: The number of participants with abnormal electrocardiogram (ECG) results is presented.
  Abnormal ECGs were considered to be those with a QTcF interval of greater than 450 msec for males and greater than 470 msec for females, or change from baseline of greater than 30 msec.
Time Frame: Part A (SAD): Screening up to Day 3
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (SAD): Placebo (Fasted) | Part A (SAD): Placebo (Fed) | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): 16 mg (Fasted) | Part A (SAD): 16 mg (Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted)
Number analyzed (Participants) | 10 | 2 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Part A (SAD): Number of Subjects With Clinically Significant Changes in Laboratory Evaluations
Description: The number of participants with clinically significant changes in any laboratory evaluations (clinical chemistry, haematology, coagulation, or urinalysis) is presented.
Time Frame: Part A (SAD): Screening up to Day 3
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (SAD): Placebo (Fasted) | Part A (SAD): Placebo (Fed) | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): 16 mg (Fasted) | Part A (SAD): 16 mg (Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted)
Number analyzed (Participants) | 10 | 2 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Part B (MAD): Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: as for outcome 5
Time Frame: Part B (MAD): Screening up to Day 14(±3)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (MAD): Placebo | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
Number analyzed (Participants) | 7 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0

9. Primary Outcome: Part B (MAD): Number of Participants With Abnormal ECG
Description: as for outcome 6
Time Frame: Part B (MAD): Screening up to Day 14(±3)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (MAD): Placebo | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
Number analyzed (Participants) | 7 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0

10. Primary Outcome: Part B (MAD): Number of Participants With Clinically Significant Changes in Laboratory Evaluations
Description: as for outcome 7
Time Frame: Part B (MAD): Screening up to Day 14(±3)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (MAD): Placebo | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
Number analyzed (Participants) | 7 | 7 | 6 | 6
Participants
  Change in leukocyte count (to above the reference range) | 0 | 0 | 0 | 1
  Change in any other evaluation | 0 | 0 | 0 | 0

11. Secondary Outcome: Part A (SAD) - Primary PK Parameters Derived From Plasma Concentration-time Profile of AQ280: Area Under the Concentration Time Curve From Time 0 Extrapolated to Infinity
Description: Primary PK parameters derived from plasma concentration-time profile of AQ280: area under the concentration time curve from time 0 extrapolated to infinity following Single Oral Dose Administration of 3, 9, 16, 48, and 60 mg AQ280 in a Fasted State and 16 mg AQ280 in a Fed State
Time Frame: Days 1, 2 and 3
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): 16 mg (Fasted) | Part A (SAD): 16 mg (Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL | 77.0 (17.2) | 318 (23.8) | 539 (35.4) | 527 (33.7) | 1860 (43.2) | 2820 (26.5)
Statistical Analysis 1: Comparison: Part A (SAD): 3 mg (Fasted) vs Part A (SAD): 9 mg (Fasted) vs Part A (SAD): 16 mg (Fasted) vs Part A (SAD): 16 mg (Fed) vs Part A (SAD): 48 mg (Fasted) vs Part A (SAD): 60 mg (Fasted); Statistical Analysis of AQ280 Primary Pharmacokinetic Endpoints to Assess Dose Proportionality of Single Oral Doses of 3 to 60 mg AQ280; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; p = 0.6358, Lack of fit 2-sided; Lack of Fit Model: ln(parameter) = intercept + slope × ln(dose) + dose + random error; Slope = 1.17, 95% CI 2-sided [1.07 to 1.27] — Between-subject geometric coefficient of variation was 30.4. Data were analyzed using a power model. ln(parameter) = intercept + slope ×ln(dose) + random error
Statistical Analysis 2: Comparison: Part A (SAD): 9 mg (Fasted) vs Part A (SAD): 16 mg (Fasted) vs Part A (SAD): 16 mg (Fed) vs Part A (SAD): 48 mg (Fasted) vs Part A (SAD): 60 mg (Fasted); Statistical Analysis of AQ280 Primary Pharmacokinetic Endpoints to Assess Dose Proportionality of Single Oral Doses of 9 to 60 mg AQ280; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; p = 0.5506, Lack of Fit 2-sided; Lack of Fit Model: ln(parameter) = intercept + slope × ln(dose) + dose + random error; Slope = 1.13, 95% CI 2-sided [0.963 to 1.31] — Between-subject geometric coefficient of variation was 32.9. Data were analyzed using a power model. ln(parameter) = intercept + slope ×ln(dose) + random error

12. Secondary Outcome: Part A (SAD) - Primary PK Parameter Derived From Plasma Concentration-time Profile of AQ280: Maximum Observed Concentration (Cmax)
Description: Part A (SAD) - Primary PK parameter derived from plasma concentration-time profile of AQ280: maximum observed concentration (Cmax) following Single Oral Dose Administration of 3, 9, 16, 48, and 60 mg AQ280 in a Fasted State and 16 mg AQ280 in a Fed State
Time Frame: Days 1, 2 and 3
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part A (SAD): 16 mg (Fasted); Part A (SAD): 16 mg (Fed): Single dose of 16 mg AQ280, fed
  AQ280: Dose form: capsule, hard Method of administration: oral
Arm/Group | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): 16 mg (Fasted) | Part A (SAD): 16 mg (Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 20.0 (16.1) | 70.1 (25.1) | 113 (16.5) | 90.8 (19.6) | 418 (40.8) | 638 (23.3)
Statistical Analysis 1: Comparison: Part A (SAD): 3 mg (Fasted) vs Part A (SAD): 9 mg (Fasted) vs Part A (SAD): 16 mg (Fasted) vs Part A (SAD): 16 mg (Fed) vs Part A (SAD): 48 mg (Fasted) vs Part A (SAD): 60 mg (Fasted); [analysis description as in outcome 11, analysis 1]; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; p = 0.3653, Lack of Fit 2-sided; Lack of Fit Model: ln(parameter) = intercept + slope × ln(dose) + dose + random error; Slope = 1.13, 95% CI 2-sided [1.04 to 1.22] — Between-subject geometric coefficient of variation was 25.7. Data were analyzed using a power model. ln(parameter) = intercept + slope ×ln(dose) + random error
Statistical Analysis 2: Comparison: Part A (SAD): 9 mg (Fasted) vs Part A (SAD): 16 mg (Fasted) vs Part A (SAD): 16 mg (Fed) vs Part A (SAD): 48 mg (Fasted) vs Part A (SAD): 60 mg (Fasted); [analysis description as in outcome 11, analysis 2]; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; p = 0.2933, Lack of Fit 2-sided; Lack of Fit Model: ln(parameter) = intercept + slope × ln(dose) + dose + random error; Slope = 1.16, 95% CI 2-sided [1.01 to 1.31] — Between-subject geometric coefficient of variation was 27.7. Data were analyzed using a power model. ln(parameter) = intercept + slope ×ln(dose) + random error

13. Secondary Outcome: Part A (SAD) - Primary PK Parameter Derived From Plasma Concentration-time Profile of the AQ280 Main Metabolite, AQ282: Area Under the Concentration Time Curve From Time 0 Extrapolated to Infinity
Description: Area under the concentration time curve from time 0 extrapolated to infinity of metabolite AQ282 following single oral dose administration of 3, 9, 16, 48, and 60 mg AQ280 in a fasted state and 16 mg AQ280 in a fed state
Time Frame: Days 1, 2 and 3
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): 16 mg (Fasted) | Part A (SAD): 16 mg (Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted)
Number analyzed (Participants) | 2 | 6 | 6 | 6 | 6 | 6
h*ng/mL | NA (NA) — Insufficient number of participants with events | 32.7 (28.2) | 43.7 (68.9) | 45.1 (66.4) | 239 (75.8) | 210 (82.0)
Statistical Analysis 1: Comparison: Part A (SAD): 3 mg (Fasted) vs Part A (SAD): 9 mg (Fasted) vs Part A (SAD): 16 mg (Fasted) vs Part A (SAD): 16 mg (Fed) vs Part A (SAD): 48 mg (Fasted) vs Part A (SAD): 60 mg (Fasted); Statistical Analysis of Metabolite AQ282 Primary Pharmacokinetic Endpoints to Assess Dose Proportionality of Single Oral Doses of 3 to 60 mg AQ280; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; p = 0.4600, Lack of Fit 2-sided; Lack of Fit Model: ln(parameter) = intercept + slope × ln(dose) + dose + random error; Slope = 1.16, 95% CI 2-sided [0.908 to 1.41] — Between-subject geometric coefficient of variation was 64.3. Data were analyzed using a power model. ln(parameter) = intercept + slope ×ln(dose) + random error
Statistical Analysis 2: Comparison: Part A (SAD): 9 mg (Fasted) vs Part A (SAD): 16 mg (Fasted) vs Part A (SAD): 16 mg (Fed) vs Part A (SAD): 48 mg (Fasted) vs Part A (SAD): 60 mg (Fasted); Statistical Analysis of Metabolite AQ282 Primary Pharmacokinetic Endpoints to Assess Dose Proportionality of Single Oral Doses of 9 to 60 mg AQ280; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; p = 0.3157, Lack of Fit 2-sided; Lack of Fit Model: ln(parameter) = intercept + slope × ln(dose) + dose + random error; Slope = 1.12, 95% CI 2-sided [0.795 to 1.45] — Between-subject geometric coefficient of variation was 65.6. Data were analyzed using a power model. ln(parameter) = intercept + slope ×ln(dose) + random error

14. Secondary Outcome: Part A (SAD) - Primary PK Parameter Derived From Plasma Concentration-time Profile of the AQ280 Main Metabolite, AQ282: Maximum Observed Concentration (Cmax)
Description: Maximum observed concentration (Cmax) of metabolite AQ282 following single oral dose administration of 3, 9, 16, 48, and 60 mg AQ280 in a fasted state and 16 mg AQ280 in a fed state
Time Frame: Days 1, 2 and 3
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): 16 mg (Fasted) | Part A (SAD): 16 mg (Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 0.722 (34.4) | 3.38 (22.4) | 3.91 (55.9) | 3.84 (62.4) | 24.4 (81.2) | 24.4 (64.8)
Statistical Analysis 1: Comparison: Part A (SAD): 3 mg (Fasted) vs Part A (SAD): 9 mg (Fasted) vs Part A (SAD): 16 mg (Fasted) vs Part A (SAD): 16 mg (Fed) vs Part A (SAD): 48 mg (Fasted) vs Part A (SAD): 60 mg (Fasted); [analysis description as in outcome 13, analysis 1]; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; p = 0.2350, Lack of fit 1-sided p-value; Lack of Fit Model: ln(parameter) = intercept + slope × ln(dose) + dose + random error; Slope = 1.20, 95% CI 2-sided [1.02 to 1.37] — Between-subject geometric coefficient of variation was 54.2. Data were analyzed using a power model. ln(parameter) = intercept + slope ×ln(dose) + random error
Statistical Analysis 2: Comparison: Part A (SAD): 9 mg (Fasted) vs Part A (SAD): 16 mg (Fasted) vs Part A (SAD): 16 mg (Fed) vs Part A (SAD): 48 mg (Fasted) vs Part A (SAD): 60 mg (Fasted); [analysis description as in outcome 13, analysis 2]; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; p = 0.1632, Lack of fit 1-sided p-value; Lack of Fit Model: ln(parameter) = intercept + slope × ln(dose) + dose + random error; Slope = 1.19, 95% CI 2-sided [0.880 to 1.50] — Between-subject geometric coefficient of variation was 58.5. Data were analyzed using a power model. ln(parameter) = intercept + slope ×ln(dose) + random error

15. Secondary Outcome: Part A (SAD) - Difference in Area Under the Concentration Time Curve From Time 0 Extrapolated to Infinity in Fasted State and in Fed State
Description: Difference in area under the concentration time curve from time 0 extrapolated to infinity derived from plasma concentration-time profile of AQ280 in fasted state and in fed state to assess the effect of food on single oral doses of 16 mg AQ280.
  The within-subject coefficient of variation is presented under the 16 mg fed results.
Time Frame: Days 1, 2 and 3
Population: Pharmacokinetic population of the 16mg fed and fasted groups in Part A. No other dose groups were assessed for food effect.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A (SAD): 16 mg (Fasted) | Part A (SAD): 16 mg (Fed)
Number analyzed (Participants) | 6 | 6
h*ng/mL | 539 (NA) — Within-subject CV of fed versus fasted is presented in the fed group results | 527 (5.66)
Statistical Analysis 1: Comparison: Part A (SAD): 16 mg (Fasted) vs Part A (SAD): 16 mg (Fed); Statistical Analysis of AQ280 Primary Pharmacokinetic Endpoints to Assess the Effect of Food on Single Oral Doses of 16 mg AQ280; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Ratio of geometric least squares mean = 0.977, 90% CI 2-sided [0.915 to 1.04] — Within-subject geometric coefficient of variation was 5.66. Data analyzed using a mixed model included treatment as a fixed effect and subject as a random effect. ln(parameter)=treatment+subject+random error, with subject fitted as a random effect

16. Secondary Outcome: Part A (SAD) - Difference in Maximum Observed Concentration (Cmax) in Fasted State and in Fed State
Description: Difference in maximum observed concentration (Cmax) derived from plasma concentration-time profile of AQ280 in fasted state and in fed state to assess the effect of food on single oral doses of 16 mg AQ280.
  The within-subject coefficient of variation is presented under the 16 mg fed results.
Time Frame: Days 1, 2 and 3
Population: as for outcome 15
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A (SAD): 16 mg (Fasted) | Part A (SAD): 16 mg (Fed)
Number analyzed (Participants) | 6 | 6
ng/mL | 113 (NA) — Within-subject CV of fed versus fasted is presented in the fed group results | 90.8 (20.5)
Statistical Analysis 1: Comparison: Part A (SAD): 16 mg (Fasted) vs Part A (SAD): 16 mg (Fed); [analysis description as in outcome 15, analysis 1]; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Ratio of geometric least squares mean = 0.805, 90% CI 2-sided [0.635 to 1.02] — Within-subject geometric coefficient of variation was 20.5. Data analyzed using a mixed model included treatment as a fixed effect and subject as a random effect. ln(parameter)=treatment+subject+random error, with subject fitted as a random effect

17. Secondary Outcome: Part B (MAD) - Primary PK Parameters Derived From Plasma Concentration-time Profile of AQ280: Accumulation Ratio (AR)
Description: Accumulation ratio (AR) AQ280 following multiple oral dose administration of 9, 27, and 60 mg AQ280 once daily for 7 consecutive days in a fasted state on Day 7.
  ARAUC = accumulation ratio based on area under the concentration-time curve over a dosing interval ARCmax = accumulation ratio based on maximum observed concentration
Time Frame: Day 1 to Day 7
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
Number analyzed (Participants) | 6 | 6 | 5
ratio
  ARAUC | 1.13 (12.0) | 1.03 (11.4) | 1.12 (5.5)
  ARCmax | 1.11 (22.7) | 0.910 (20.0) | 1.12 (13.1)

18. Secondary Outcome: Part B (MAD) - Primary PK Parameters Derived From Plasma Concentration-time Profile of AQ280: Area Under the Concentration Time Curve Over a Dosing Interval
Description: Area under the concentration time curve over a dosing interval (AUCτ) following single oral administration of 9, 27, and 60 mg AQ280 in a fasted state (Day 1) and after multiple oral dose administration of 9, 27, and 60 mg AQ280 once daily for 7 consecutive days in a fasted state (Day 7).
Time Frame: Day 1 and Day 7
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
Number analyzed (Participants) | 7 | 6 | 6
h*ng/mL
  Day 1 | 300 (28.9) | 978 (29.8) | 2910 (36.8)
  Day 7: number analyzed (Participants) | 6 | 6 | 5
  Day 7 | 345 (26.1) | 1000 (21.7) | 3150 (36.4)
Statistical Analysis 1: Comparison: Part B (MAD): 9 mg vs Part B (MAD): 27 mg vs Part B (MAD): 60 mg; Statistical Analysis of AQ280 Primary Pharmacokinetic Endpoints to Assess Dose Proportionality of Multiple Oral Doses of 9 to 60 mg AQ280 QD for 7 Consecutive Days in a Fasted State; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; p = 0.1558, Lack of fit 2-sided; Lack of Fit Model: ln(parameter) = intercept + slope × ln(dose) + dose + random error; Slope = 1.15, 95% CI 2-sided [0.954 to 1.34] — Between-subject geometric coefficient of variation was 28.0. Data were analyzed using a power model. ln(parameter) = intercept + slope ×ln(dose) + random error

19. Secondary Outcome: Part B (MAD) - Primary PK Parameters Derived From Plasma Concentration-time Profile of AQ280: Maximum Observed Concentration (Cmax)
Description: Maximum observed concentration (Cmax) following single oral administration of 9, 27, and 60 mg AQ280 in a fasted state (Day 1) and after multiple oral dose administration of 9, 27, and 60 mg AQ280 once daily for 7 consecutive days in a fasted state (Day 7).
Time Frame: Day 1 and Day 7
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
Number analyzed (Participants) | 7 | 6 | 6
ng/mL
  Day 1 | 64.5 (30.1) | 248 (24.3) | 560 (32.1)
  Day 7: number analyzed (Participants) | 6 | 6 | 5
  Day 7 | 72.0 (23.0) | 226 (20.5) | 590 (28.8)
Statistical Analysis 1: Comparison: Part B (MAD): 9 mg vs Part B (MAD): 27 mg vs Part B (MAD): 60 mg; [analysis description as in outcome 18, analysis 1]; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; p = 0.5458, Lack of Fit 2-sided model; Lack of Fit Model: ln(parameter) = intercept + slope × ln(dose) + dose + random error; Slope = 1.10, 95% CI 2-sided [0.946 to 1.26] — Between-subject geometric coefficient of variation was 24.0. Data were analyzed using a power model. ln(parameter) = intercept + slope ×ln(dose) + random error

20. Secondary Outcome: Part B (MAD) - Primary PK Parameter Derived From Plasma Concentration-time Profile of the AQ280 Main Metabolite, AQ282: Area Under the Concentration Time Curve Over a Dosing Interval (AUCτ)
Description: Area under the concentration time curve over a dosing interval (AUCτ) of metabolite AQ282 following single oral dose administration of 9, 27, and 60 mg AQ280 in a fasted state (Day 1) and multiple oral dose administration of 9, 27, and 60 mg AQ280 once daily for 7 consecutive days in a fasted state (Day 7).
Time Frame: Day 1 and Day 7
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
Number analyzed (Participants) | 7 | 6 | 6
h*ng/mL
  Day 1 | 31.3 (33.7) | 121 (43.1) | 217 (44.4)
  Day 7: number analyzed (Participants) | 6 | 6 | 5
  Day 7 | 37.0 (29.7) | 123 (61.0) | 214 (71.6)
Statistical Analysis 1: Comparison: Part B (MAD): 9 mg vs Part B (MAD): 27 mg vs Part B (MAD): 60 mg; Statistical Analysis of Metabolite AQ282 Primary Pharmacokinetic Endpoints to Assess Dose Proportionality of Multiple Oral Doses of 9 to 60 mg AQ280 once daily for 7 Consecutive Days in a Fasted State; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; p = 0.4856, Lack of fit 2-sided — Lack of Fit Model: ln(parameter) = intercept + slope × ln(dose) + dose + random error; Slope = 0.941, 95% CI 2-sided [0.602 to 1.28] — Between-subject geometric coefficient of variation was 54.7. Data were analyzed using a power model. ln(parameter) = intercept + slope ×ln(dose) + random error

21. Secondary Outcome: Part B (MAD) - Primary PK Parameter Derived From Plasma Concentration-time Profile of the AQ280 Main Metabolite, AQ282: Maximum Observed Concentration (Cmax)
Description: Maximum observed concentration (Cmax) of metabolite AQ282 following single oral dose administration of 9, 27, and 60 mg AQ280 in a fasted state (Day 1) and multiple oral dose administration of 9, 27, and 60 mg AQ280 once daily for 7 consecutive days in a fasted state (Day 7).
Time Frame: Day 1 and Day 7
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
Number analyzed (Participants) | 7 | 6 | 6
ng/mL
  Day 1 | 3.37 (25.3) | 15.6 (35.1) | 24.6 (35.9)
  Day 7: number analyzed (Participants) | 6 | 6 | 5
  Day 7 | 3.59 (15.9) | 14.2 (53.0) | 21.3 (61.1)
Statistical Analysis 1: Comparison: Part B (MAD): 9 mg vs Part B (MAD): 27 mg vs Part B (MAD): 60 mg; [analysis description as in outcome 20, analysis 1]; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; p = 0.1455, Lack of fit 2-sided; Lack of Fit Model: ln(parameter) = intercept + slope × ln(dose) + dose + random error; Slope = 0.971, 95% CI 2-sided [0.666 to 1.28] — Between-subject geometric coefficient of variation was 45.5. Data were analyzed using a power model. ln(parameter) = intercept + slope ×ln(dose) + random error

ADVERSE EVENTS:
Time Frame: Part A: up to 7 weeks, from screening up to safety follow up Part B: up to 8 weeks, from screening up to safety follow up
Description: The 'Part A (SAD): Placebo (Fasted)' cohort includes the 8 participants in the fasted only cohort as well as any AEs experienced by the 2 participants in the 'Part A (SAD): Placebo (Fasted/Fed)' cohort whilst in the fasting during Treatment Period 1. Any AEs experienced by these 2 participants during Treatment Period 2 (ie, the fed stage) only are listed separately under the cohort 'Part A (SAD): Placebo (Fed).
Arm/Group | Part A (SAD): Placebo (Fasted) | Part A (SAD): Placebo (Fed) | Part A (SAD): 3 mg (Fasted) | Part A (SAD): 9 mg (Fasted) | Part A (SAD): 16 mg (Fasted) | Part A (SAD): 16 mg (Fed) | Part A (SAD): 48 mg (Fasted) | Part A (SAD): 60 mg (Fasted) | Part B (MAD): Placebo | Part B (MAD): 9 mg | Part B (MAD): 27 mg | Part B (MAD): 60 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/7 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/7 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/10 | 0/2 | 1/6 | 2/6 | 1/6 | 2/6 | 0/6 | 1/6 | 3/7 | 3/7 | 3/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (SAD): Placebo (Fasted) (N=10) | Part A (SAD): Placebo (Fed) (N=2) | Part A (SAD): 3 mg (Fasted) (N=6) | Part A (SAD): 9 mg (Fasted) (N=6) | Part A (SAD): 16 mg (Fasted) (N=6) | Part A (SAD): 16 mg (Fed) (N=6) | Part A (SAD): 48 mg (Fasted) (N=6) | Part A (SAD): 60 mg (Fasted) (N=6) | Part B (MAD): Placebo (N=7) | Part B (MAD): 9 mg (N=7) | Part B (MAD): 27 mg (N=6) | Part B (MAD): 60 mg (N=6)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. If foreseen, the PI agrees to submit all manuscripts or abstracts to the sponsor before submission.

The sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/79/NCT05485779/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT05485779/SAP_001.pdf